CLINICAL TRIAL: NCT02549898
Title: Investigation of Vascular Inflammation in Migraine Without Aura Using Molecular Nano-imaging and Black Blood Imaging MRI
Brief Title: Investigation of Vascular Inflammation in Migraine Using Molecular Nano-imaging and Black Blood Imaging MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Sabrina Khan, Medical Doctor and PhD student, Danish Headache Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-15005669
Record Dates: First submitted 2015-07-31; First posted 2015-09-15 (Estimated); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Migraine Headache; Migraine Without Aura
MeSH Terms: conditions — Migraine Disorders; Migraine without Aura | interventions — Ferrosoferric Oxide; Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vascular inflammation (Experimental): Subjects with habitual unilateral migraine without aura, undergo a baseline MRI scan, undergo pharmacological induction of a migraine attack, and subsequently are MRI scanned prior to (BBI-MRI) and after Feraheme infusion (USPIO-MRI ).
  Interventions: Drug: Feraheme; Drug: Cilostazol; Other: USPIO-MRI; Other: BBI-MRI
- Effect of sumatriptan (Experimental): Subjects with habitual unilateral migraine without aura, undergo a baseline MRI scan and then undergo pharmacological induction of a migraine attack. Sumatriptan is given and subjects subsequently undergo MRI scans prior to (BBI-MRI) and after Feraheme infusion (USPIO-MRI).
  Interventions: Drug: Feraheme; Drug: Cilostazol; Other: USPIO-MRI; Other: BBI-MRI
- Pilot w/o cilostazol (Experimental): Subjects without habitual unilateral migraine without aura undergo a baseline MRI scan. Subjects are then MRI scanned prior to (BBI-MRI) and after Feraheme infusion (USPIO-MRI).
  Interventions: Drug: Feraheme; Other: USPIO-MRI; Other: BBI-MRI
- Pilot w/ cilostazol (Experimental): Subjects without habitual unilateral migraine without aura undergo a baseline MRI scan and then receive cilostazol. Subjects are then MRI scanned prior (BBI-MRI) to and after Feraheme infusion (USPIO-MRI).
  Interventions: Drug: Feraheme; Drug: Cilostazol; Other: USPIO-MRI; Other: BBI-MRI

INTERVENTIONS:
Drug: Feraheme — Feraheme is an USPIO agent, which will be applied as a contrast agent to visualize vascular inflammation in unilateral migraine without aura.
  Other Names: Ferumoxytol
Drug: Cilostazol — Cilostazol will be applied to provoke migraine attacks in migraineurs
  Other Names: Pletal
  Arms: Effect of sumatriptan; Pilot w/ cilostazol; Vascular inflammation
Other: USPIO-MRI — USPIO-MRI scans will be performed in order to assess possible vascular inflammation associated with migraine attacks.
Other: BBI-MRI — Black blood MRI scans will be performed in order to asses changes in vessel wall thickness due to possible vascular inflammation associated with migraine attacks.

SUMMARY:
The investigators aim to investigate inflammation of cranial and meningeal arteries during pharmacologically induced migraine attacks, using ultrasmall superparamagnetic iron oxide (USPIO) nanoparticles and black blood imaging (BBI) MRI.

DETAILED DESCRIPTION:
Migraine is the most common neurological disorder, ranked as the 7th most debilitating disease worldwide by the WHO. While much research has been and continues to be conducted to illuminate the enigma of migraine pathophysiology, key aspects still remain a conundrum. Specifically, the process of headache generation is perhaps the most complex and debated part of migraine pathophysiology. The vascular hypothesis of migraine has traditionally focused on the simple dilatation of cranial arteries. However, a possible contribution of perivascular pain sensitive structures should also be considered, as aseptic inflammation of the arterial walls and perivascular space may activate afferent nerve endings. Interestingly, giant cell arteritis caused by aseptic arterial wall inflammation may present clinically as localized headache with migraine-like features (i.e. throbbing pain, localized in the temporal region, and allodynia).

The primary trigeminal nociceptor is the first integral part of the headache-generating pathway. Animal models of migraine have suggested that activation and sensitization of perivascular trigeminal nociceptors caused by inflammatory substances may explain head pain in migraine. However, there is no human evidence to date to suggest perivascular and arterial wall inflammation as a source of pain in migraine.

The investigators hypothesize that unilateral migraine without aura is associated with ipsilateral inflammation of the cranial arteries and meninges. The investigators also suggest that sumatriptan inhibits this perivascular inflammation. To test the hypotheses the investigators will perform MRI scans on subjects with provoked migraine attacks, using two different methods to visualize perivascular inflammation: USPIO-MRI, using iron-oxide nanoparticles as contrast agent, and BBI MRI.

To pharmacologically induce migraine headache in the study subjects, the investigators will use the drug cilostazol, which is a phosphodiesterase 3 inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Subject has migraine without aura according to criteria of the International Headache Society (IHS)
* Subject has unilateral migraine 70% of the time
* Migraine can be pharmacologically provoked in the subject using cilostazol.
* Subject is on birth control
* Subject has no other medical history

Exclusion Criteria:

* Subject suffers from bilateral migraine
* Subject suffers from migraine with aura
* Subject suffers from other primary headaches as specified by IHS criteria
* Pregnant or breast feeding subjects
* Subjects with contraindications for undergoing MRI scans
* Any known drug allergy
* Any signs or disorders of iron overload, including but not limited to hemosiderosis and porphyria cutanea tarda

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2015-08; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change in USPIO uptake during attacks of unilateral migraine without aura compared to baseline | 34 hours
  On the first study day, migraine is induced with cilostazol, and intravenous infusion of Feraheme (USPIO) is delivered. On the second study day, USPIO-MRI is performed.
Change in arterial wall thickness during attacks of unilateral migraine without aura compared to baseline | 6 hours
  On the first study day, migraine is induced with cilostazol, and 4 hours after cilostazol ingestion, BBI-MRI is performed.
Change in arterial circumference as a proxy measure for vascular inflammation during attacks of unilateral migraine without aura compared to baseline | 34 hours
  On the first study day, migraine is induced with cilostazol, and at 4 hours and 28 hours after cilostazol ingestion, MR angiography is performed.
Change in USPIO uptake during attacks of unilateral migraine without aura before and after sumatriptan | 36 hours
  On the first study day, migraine is induced with cilostazol and subsequently treated with sumatriptan. Intravenous infusion of Feraheme (USPIO) is delivered, and on the second study day, USPIO-MRI is performed.
Change in arterial wall thickness during attacks of unilateral migraine without aura before and after sumatriptan | 7 hours
  On the first study day, migraine is induced with cilostazol, and 4 hours after cilostazol ingestion, BBI-MRI is performed. Subjects are treated with sumatriptan, and BBI-MRI is repeated.
Change in arterial circumference as a proxy measure for vascular inflammation during unilateral attacks of migraine without aura before and after sumatriptan | 36 hours
  On the first study day, migraine is induced with cilostazol, and 4 hours after cilostazol, MR angiography is performed. Subjects are treated with sumatriptan, and MR angiography is repeated. 28 hours after cilostazol ingestion, MR angiography is performed again.

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Khan, MD, Principal Investigator — Danish Headache Center
Locations (1):
- Rigshospitalet Glostrup, Glostrup Municipality, Denmark

REFERENCES:
- [Derived] Khan S, Amin FM, Fliedner FP, Christensen CE, Tolnai D, Younis S, Olinger ACR, Birgens H, Daldrup-Link H, Kjaer A, Larsson HBW, Lindberg U, Ashina M. Investigating macrophage-mediated inflammation in migraine using ultrasmall superparamagnetic iron oxide-enhanced 3T magnetic resonance imaging. Cephalalgia. 2019 Oct;39(11):1407-1420. doi: 10.1177/0333102419848122. Epub 2019 May 19. PMID 31104505